CLINICAL TRIAL: NCT03753425
Title: Colonoscopy With Low Volume bowEl prepAration in iNflammatory Bowel Diseases
Brief Title: National Multicentric Observatory of Low Bowel Preparations in Patients With IBD
Acronym: CLEAN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/310
Record Dates: First submitted 2017-10-19; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2017-10

CONDITIONS: Patient With an Indication of Colonoscopy for Inflammatory Bowel Disease
Keywords: Inflammatory bowel disease; colonoscopy; bowel preparations
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- PEG4L, four liters polyethylene glycol: PEG4L, four liters polyethylene glycol
- PEG2L, two liters polyethylene glycol with ascorbic acid: PEG2L, two liters polyethylene glycol with ascorbic acid
- Pico, sodium picosulfate: Pico, sodium picosulfate
- NaP, sodium phosphate: NaP, sodium phosphate
- MPS, sodium, magnesium and potassium sulphates: MPS, sodium, magnesium and potassium sulphates
  Interventions: Procedure: Low volume bowel preparation in inflammatory bowel diseases

INTERVENTIONS:
Procedure: Low volume bowel preparation in inflammatory bowel diseases — Low volume bowel preparation in inflammatory bowel diseases
  Other Names: Preparation in inflammatory bowel diseases given to patients before a coloscopy
  Groups: MPS, sodium, magnesium and potassium sulphates

SUMMARY:
National multicentric observatory of low bowel preparations in patients with IBD

DETAILED DESCRIPTION:
Prospective french multicentre observational study, during one month: from March 6th to April 6th 2017, under the auspice of the IBD group of the Société Française d'Endoscopie Digestive- SFED. All French gastroenterologists in charge of IBD patients in public or private endoscopy centers were reached out through various professional and scientific associations to participate in the study via e-mail, web sites, and national congresses. Investigators were asked to prescribe the bowel preparation independently from the study, as per their usual habits. The achievement of low residue diet, the split and the timing of the preparation were left free to the investigator according to local protocols.

Data recording The physicians participating in the study completed data on an online questionnaire via an internet-based tool (CleanWeb software, hosted by Besançon university hospital research center) or through a questionnaire sheet. The questionnaire included a medical record and a self-reported patient questionnaire. The medical record included physicians and centers characteristics, patient's demographics, disease characteristics, modality of bowel preparation (diet, split dose, type of bowel preparation, delay before colonoscopy), and colonoscopy findings and outcomes. Patients self-administered questionnaires assessed preparation tolerability by symptoms and satisfaction recording.

Clinical endpoints The efficacy of the preparation was evaluated by the Boston's score (efficacy was defined as a Boston's score was ≥ 7 without any segment <2)23, the rate of caecal or anastomosis intubation and the necessity or not to repeat the colonoscopy.

The tolerance was evaluated by the quantity of preparation actually absorbed by the patient, (quantity of active preparation and quantity of clear liquid), patients and investigators visual analogue scale evaluation of tolerance (VAS), a self-administered validated bowel-preparation tolerability questionnaire 24 and by the patients' wish to take the same preparation for the next colonoscopy.

Safety data: adverse events were collected per preparation and per endoscopic procedure, at 24 hours and 30 days later. A special focus was made on aphtoid lesions as they were previously reported as adverse preparation-induced mucosal lesions possibly associated with some solutions.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-75 years,
* symptoms of IBD for at least 3 month,
* inidcation of colonoscopy independent from the study.

Exclusion Criteria:

* Congestive heart failure,
* severe renal failure,
* gastro intestinal symptomatic obstruction or occlusive bowel stenosis (a non-occlusive stenosis was not an exclusion criterion),
* severe acute colitis,
* severe dehydration or electrolyte disturbances,
* patient's refusal to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication of colonoscopy independent from the study
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-06-03 (Actual)

PRIMARY OUTCOMES:
Boston Score | 30 days
  According to the rate of complete colonoscopy (caecal intubation); and according to the need to reschedule the examination

SECONDARY OUTCOMES:
tolerance: visual analogue scale | 30 days
  visual analogue scale
adverse events per procedure | 30 days
  fever, bowel perforation, bleeding, inhalation, hospitalisation, disease flare

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hosptalier Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No